CLINICAL TRIAL: NCT01489449
Title: Bare Metal Stent Versus Drug Coated Balloon With Provisional Stenting in Non-ST-Elevation Myocardial Infarction
Acronym: PEPCADNSTEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEPCAD NSTEMI
Record Dates: First submitted 2011-11-27; First posted 2011-12-09 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Coronary Heart Disease; NSTEMI
Keywords: drug coated balloon; NSTEMI
MeSH Terms: conditions — Coronary Disease; Non-ST Elevated Myocardial Infarction | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent (Placebo Comparator): Stent Implantation (DES or BMS), no further treatment
  Interventions: Device: Stent
- DCB (Active Comparator): "DEBonly" strategy: treatment with drug coated balloon, additional spot-stenting in case of severe dissection
  Interventions: Combination Product: SeQuent(R) Please coated balloon

INTERVENTIONS:
Device: Stent — bare metal stent implantation, any bare metal stent is allowed from different companies
  Arms: Stent
Combination Product: SeQuent(R) Please coated balloon — Angioplasty with Drug coated balloon (DCB)
  Other Names: SeQuent(R) Please
  Arms: DCB

SUMMARY:
The aim of the present trial is to assess the efficacy of the standalone use of SeQuent(R) Please coated balloon compared to a bare metal stent (BMS) in patients with NSTEMI.

DETAILED DESCRIPTION:
The aim of the present trial is to assess the efficacy of the standalone use of SeQuent(R) Please coated balloon compared to a bare metal stent (BMS) in patients with NSTEMI. Primary efficacy endpoint will be MACE (cardiac mortality, reinfarction, and target lesion revascularization) after 9 months.

ELIGIBILITY:
Inclusion Criteria:

* NSTEMI with
* Ischemic symptoms (angina pectoris) > 30 minutes
* Last symptoms within 72 hours before randomization
* Positive cardiac troponin T, I, or hs-Troponin above 99th percentile
* age > 18 years
* Identifiable culprit lesion without angiographic evidence of large thrombus with intended early PCI (treatment of up to two lesions allowed)

Exclusion Criteria:

* Cardiogenic shock
* ST-elevation myocardial infarction
* No identifiable culprit lesion, Indication for acute bypass surgery
* Comorbidity with limited life expectancy < 9-12 months
* Contraindication for treatment with heparin, ASA and thienopyridines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
MACE | 9 months
  MACE means the occurence of cardiac death, reinfarction, or target lesion revascularization

SECONDARY OUTCOMES:
Stent thrombosis (ARC | 9 months, 3 years, 5 years
Mortality (cardiac and non-cardiac) | 9 months, 3 years, 5 years
Reinfarction | 9 months, 3 years, 5 years
target lesion revascularization | 9 months, 3 years, 5 years
target vessel revascularization | 9 months, 3 years, 5 years
any revascularization | 9 months, 3 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes
Locations (1):
- Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Derived] Scheller B, Ohlow MA, Ewen S, Kische S, Rudolph TK, Clever YP, Wagner A, Richter S, El-Garhy M, Bohm M, Degenhardt R, Mahfoud F, Lauer B. Bare metal or drug-eluting stent versus drug-coated balloon in non-ST-elevation myocardial infarction: the randomised PEPCAD NSTEMI trial. EuroIntervention. 2020 Apr 17;15(17):1527-1533. doi: 10.4244/EIJ-D-19-00723. PMID 31659986